CLINICAL TRIAL: NCT01148043
Title: Pharmacological Treatment In Osteoarthritis
Acronym: FABIO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maasstad Hospital (Other)
Responsible Party: Principal Investigator, WeiChing Lee, pharmacist, Maasstad Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL32030.101.10
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Hydroxychloroquine; Cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: cellulose
- Hydroxychloroquine (Experimental)
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — 200 mg capsule, 2 capsules QD for 24 weeks.
  Other Names: Plaquenil
  Arms: Hydroxychloroquine
Drug: cellulose — capsule, 2 capsules QD for 24 weeks
  Other Names: placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of hydroxychloroquine in hand osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis is the most common joint disease, most frequently involving the hands, resulting in pain, stiffness and loss of hand function. At present, there is no option to prevent the onset or the progression of hand osteoarthritis (OA). It is believed that inflammation plays an important role in the pathogenesis of OA and that anti-inflammatory drugs might be an effective treatment for OA. Anti-malarial agents like chloroquine and hydroxychloroquine are potential anti-inflammatory drugs and hydroxychloroquine has already proven to be an effective suppressor of inflammation in rheumatoid arthritis. Several previous studies with hydroxychloroquine in hand OA also showed a possible effect on pain and inflammation, but these studies were mostly retrospective with a small number of patients. This is the first prospective, randomised, placebo-controlled study to determine the effect of hydroxychloroquine in hand osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years
* Primary hand OA according to the ACR classification
* Heberden or Bouchard nodule or Kellgren-Lawrence grade 1, 2 or 3 changes in ≥ 2 symptomatic joints
* Pain in the dominant hand ≥ 12 months
* Use of an NSAID for ≥ 1 episode of pain
* Written informed consent

Exclusion Criteria:

* Secondary hand OA, e.g. haemochromatoses, rheumatoid arthritis, posttraumatic
* Kellgren-Lawrence grade 4 OA
* Use of hydroxychloroquine within 3 months before entering the study
* Use of NSAIDs or corticosteroids within 7 days before entering the study
* Retinopathy
* Myasthenia gravis
* Known allergy or hypersensitivity for hydroxychloroquine

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-07; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Pain intensity measured by 100 mm Visual Analog Scale (VAS) | 24 weeks

SECONDARY OUTCOMES:
Hand function measured by Arthritis Impact Measurement Scales 2 short form (AIMS2-SF) and Australian/Canadian Osteoarthritis Hand Index (AUSCAN) | 6, 12 and 24 weeks
Pain intensity measured by 100 mm VAS | 6, 12 weeks
Radiological progression measured by the anatomical lesion progression system from Verbruggen et al. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Natalja M Basoski, MD, Principal Investigator — Maasstad Hospital
Locations (6):
- Netherlands (6):
  - Admiraal de Ruyter Hospital, Goes
  - Maasstad Hospital, Rotterdam
  - Erasmus Medical Center, Rotterdam
  - Sint Franciscus Gasthuis, Rotterdam
  - Vlietland Hospital, Schiedam
  - ZorgSaam Zeeuws-Vlaanderen, Terneuzen

REFERENCES:
- [Derived] Lee W, Ruijgrok L, Boxma-de Klerk B, Kok MR, Kloppenburg M, Gerards A, Huisman M, Hazes M, de Sonnaville P, Grillet B, Weel A, Basoski N. Efficacy of Hydroxychloroquine in Hand Osteoarthritis: A Randomized, Double-Blind, Placebo-Controlled Trial. Arthritis Care Res (Hoboken). 2018 Sep;70(9):1320-1325. doi: 10.1002/acr.23471. Epub 2018 Aug 12. PMID 29125901